CLINICAL TRIAL: NCT01959178
Title: A Study to Evaluate a Mid Add Multi-Focal Soft Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 825E
Record Dates: First submitted 2013-10-08; First posted 2013-10-09 (Estimated); Results first posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LD127025 MF (Experimental): Mid add daily disposable soft contact lens worn on a daily wear basis for 1 week.
  Interventions: Device: LD127025 MF; Device: Air Optix Aqua MF
- Air Optix Aqua MF (Active Comparator): Medium add daily disposable soft contact lens worn on a daily wear basis for one week.
  Interventions: Device: LD127025 MF; Device: Air Optix Aqua MF

INTERVENTIONS:
Device: LD127025 MF — At Visit 1, one-half of the subjects will be randomized to receive the investigational soft contact lens, after approximately one week of wearing the first lens type, the subjects will return for the 1-Week Crossover Visit (Visit 2) for an exam, and to determine if the subject remains eligible to continue in the next phase of the study with the control soft contact lens.
Device: Air Optix Aqua MF — At Visit 1, one-half of the subjects will be randomized to receive the control soft contact lens, after approximately one week of wearing the first lens type, the subjects will return for the 1-Week Crossover Visit (Visit 2) for an exam, and to determine if the subject remains eligible to continue in the next phase of the study with the investigational soft contact lens.

SUMMARY:
This study is to evaluate the product performance of the investigational LD127025 MF mid add soft contact lens compared to CIBA Vision's Air Optix Aqua MF MED add soft contact lenses when used among currently adapted soft contact lens wearers.

ELIGIBILITY:
Inclusion Criteria

* Have physiologically normal anterior segments not exhibiting biomicroscopy findings Grade 2 or greater and/or presence of infiltrates.
* Be adapted wearers of soft contact lenses, wear a lens in each eye, and each lens must be of the same manufacture and brand.
* Be correctable through spherocylindrical refraction to 42 letters (0.1 logMAR) or better (distance, high contrast) in each eye.
* Require contact lens correction from -5.00 D to +3.00 D in each eye.
* Be Presbyopic and require near add correction from +1.00 D to +1.75 D in each eye.
* Be an adapted monovision soft contact lens wearer or multifocal soft contact lens wearer or an adapted spherical soft contact lens wearer who also uses spectacles for near vision correction.
* Be willing to use a lens care system as required by the lens replacement schedule.
* Has a distance spherical equivalent refraction between -5.50 D and +3.00 D.

Exclusion Criteria:

* Not correctable to 32 letters (0.3 logMAR) in each eye with soft spherical contact lenses.
* Participated in any drug or device clinical investigation (within 14 days) prior to entry into this study and/or during the period of study participation.
* Women of childbearing potential if one of the following: pregnant, plans to become pregnant during study, is breast-feeding.
* Any Grade 2 or greater finding during the slit lamp examination. Subjects with corneal infiltrates of ANY GRADE are not eligible.
* Any scar or neovascularization within the central 4mm of the cornea. Subjects with minor peripheral corneal scarring (that does not extend into the central area), that in the Investigator's judgment, does not interfere with contact lens wear, are eligible for this study.
* Any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.
* Anisometropia (spherical equivalent) of greater than 2.00 D.
* Aphakic.
* Amblyopic.
* Allergic to any component in the study care products.
* Meet any of the following criteria:
* Ophthalmologist, OD, Optician, Ophthalmologist's Assistant/Technician
* employee of a market research firm
* employee of manufacturer of contact lens or contact lens care products
* Ocular astigmatism of greater than 1.00 D in either eye.
* Have had any corneal surgery (ie, refractive surgery).
* Toric contact lens wearer.
* Have worn gas permeable (GP) contact lenses within the last 30 days or PMMA lenses within the last 3 months.
* Have an active ocular disease or are using any ocular medication.
* Have any systemic disease currently affecting ocular health or which, in the Investigator's opinion, may have an effect on ocular health during the course of the study.
* Using any systemic medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Stefffen, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Incorporated, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 146 participants (292 eyes) were enrolled in this study. One-half of the participants were randomized to receive the investigational lens, and the other half to the control lens. After one week, the participant crossed over to the second lens type for one week.
Groups:
- LD127025 MF Then Air Optix Aqua MF: LD127025 MF and then Air Optix Aqua MF after 1 week
- Air Optix Aqua MF Then LD127025 MF: Air Optix Aqua MF and then LD127025 MF after 1 week
Period: Overall Study
Arm/Group | LD127025 MF Then Air Optix Aqua MF | Air Optix Aqua MF Then LD127025 MF
Started | 73 | 73
Completed | 71 | 71
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Population: Demographics were reported for all eligible, dispensed participants. There was one participant that was not eligible for the study, and thus was excluded.
Groups:
- Overall Enrolled: Overall participants enrolled.
Arm/Group | Overall Enrolled
Number analyzed (Participants) | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Mean Visual Acuity
Description: Visual acuity was assessed by distance high contrast logarithm of the minimum angle of resolution (logMAR).
Time Frame: At 1 Week follow up
Population: Eligible, dispensed eyes assessed for visual acuity are included in the analysis population.
Measure: Least Squares Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | LD127025 MF | Air Optix Aqua MF
Number analyzed (Participants) | 143 | 144
Number analyzed (eyes) | 286 | 288
logMAR | -0.026 (0.070) | 0.008 (0.078)

2. Secondary Outcome: Symptoms/Complaints
Description: Symptoms/complaints were assessed on a scale from 0 to 100, with 0 denoting unfavorable symptoms/complaints.
Time Frame: At 1 Week follow up
Population: Eligible, dispensed eyes assessed for symptoms/complaints are included in the analysis population.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | LD127025 MF | Air Optix Aqua MF
Number analyzed (Participants) | 143 | 141
Number analyzed (eyes) | 286 | 282
score on a scale
  Burning/stinging upon insertion | 96.1 (9.8) | 93.4 (11.8)
  Comfort upon insertion | 95.4 (8.3) | 91.4 (12.6)
  Comfort at end of day | 83.7 (19.5) | 79.9 (20.7)
  Overall comfort | 88.3 (16.4) | 84.6 (17.4)
  Ease of handling/insertion | 92.3 (13.3) | 93.5 (9.6)
  Ease of handling/removal | 89.3 (16.5) | 93.6 (9.7)
  Dryness | 86.1 (18.2) | 85.6 (16.9)
  Itchiness | 94.4 (10.3) | 90.2 (15.1)
  Redness | 95.3 (7.6) | 91.0 (13.9)
  Overall impression | 84.1 (19.7) | 83.3 (19.9)
  Distance vision | 91.0 (16.1) | 82.0 (21.1)
  Vision at intermediate distance | 80.8 (21.8) | 84.4 (16.3)
  Vision at near distance | 60.1 (28.6) | 76.1 (22.6)
  Overall vision | 74.0 (23.0) | 79.5 (19.9)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Adverse events were not coded. Therefore, source vocabulary is not applicable. Safety data were reported for all eligible, dispensed participants. There was one participant that was not eligible for the study, and thus was excluded.
Arm/Group | LD127025 MF | Air Optix Aqua MF
Serious Adverse Events (participants affected / at risk) | 0/145 | 0/145
Other Adverse Events (participants affected / at risk) | 0/145 | 0/145

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.